CLINICAL TRIAL: NCT03798470
Title: FAVOR Opioid Recovery Coaching Evaluation
Acronym: FORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: FAVOR (Faces and Voices of Recovery) OF GREENVILLE (Unknown); South Carolina Department of Alcohol and Other Drug Abuse Services (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00073004
Record Dates: First submitted 2018-12-24; First posted 2019-01-10 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Opiate Abuse; Opiate Overdose; Opioid-use Disorder
Keywords: opioid; overdose
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort (Experimental): Intervention with FAVOR peer recovery coaching. Patients identified in the ED as opioid overdose and enrolled in the current study.
  Interventions: Behavioral: Peer Addiction Counseling

INTERVENTIONS:
Behavioral: Peer Addiction Counseling — After identification, a 24/7 on-call FRC was paged and met with the patient in the ED. The patients were offered recovery services at the bedside by the FRC. The research team members offered voluntary participation and obtained informed consent to enrolling a longitudinal study looking into the success of his intervention. Patients did not need to participate to be eligible for counseling and resources from AVOR. The FRCs counselled and engaged the patient along with the family to offer a variety of services including active recovery coaching, group treatment modalities, family support services and transportation. After he initial encounter in the ED, the FAVOR team re-engaged the participant by phone or in person the next day and gradually increasing intervals thereafter.
  Other Names: FAVOR counseling

SUMMARY:
The Emergency Department (ED) is an ideal location to identify patients in need of treatment for opioid addiction. A local non-profit community-based addiction recovery program, Faces and Voices of Recovery (FAVOR) utilizes a peer recovery coaching model applied to substance use disorders by identifying, training, credentialing and supervising individuals who have been in recovery for at least 2 years.

These peer recovery coaches become the primary workforce in this community-based model. FAVOR provides no-cost comprehensive services for addiction recovery. The investigators hypothesized that having FAVOR Recovery Coaches (FRC) evaluate patients during an ED visit for opioid overdose would result in a high degree of engagement from the patients and serve as an opportunity to begin treatment for addiction.

DETAILED DESCRIPTION:
The Emergency Department (ED) is an ideal location to identify patients in need of treatment for opioid addiction. A local non-profit community-based addiction recovery program, Faces and Voices of Recovery (FAVOR) utilizes a peer recovery coaching model applied to substance use disorders by identifying, training, credentialing and supervising individuals who have been in recovery for at least 2 years.These peer recovery coaches become the primary workforce in this community-based model. FAVOR provides no-cost comprehensive services for addiction recovery. The investigators hypothesized that having FAVOR Recovery Coaches (FRC) evaluate patients during an ED visit for opioid overdose would result in a high degree of engagement from the patients and serve as an opportunity to begin treatment for addiction.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the ED with opioid overdose or withdrawal

Exclusion Criteria:

* Age <18
* Known pregnant female
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with active involvement in recovery | One year
  Defined as: Patients who have had phone, email, or in-person contact with their FAVOR recovery coach after discharge from the Emergency Department.

SECONDARY OUTCOMES:
All-cause Mortality | One year
  Number of participants with death from any cause within the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carey, MD, Principal Investigator — Greenville Health System Emergency Medicine
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The data would be de-identified if shared.